CLINICAL TRIAL: NCT01248286
Title: Effect of Whole Grain Diet on Insulin Sensitivity, Advanced Glycation End Products and Inflammatory Markers in Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 10-0924; 10-0924 0001 01 ME (Other: Mount Sinai Grants and Contract Office)
Record Dates: First submitted 2010-11-17; First posted 2010-11-25 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes; Prediabetes
Keywords: Diabetes; Prediabetes; Prevention; Whole grain; Advanced glycation end products; Insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole grain rice (Experimental)
  Interventions: Other: Whole grain rice
- Refined grain rice (Active Comparator)
  Interventions: Other: Refined grain rice

INTERVENTIONS:
Other: Whole grain rice — Whole grain rice arm (treatment arm): Subjects will be provided a supply of whole grain rice and will be asked to prepare rice items in their meal with the provided whole grain rice while participating in the study
  Arms: Whole grain rice
Other: Refined grain rice — Refined grain rice arm (control arm): Subjects will be provided a supply of refined grain rice and will be asked to prepare rice items in their meal with the provided refined grain rice while participating in the study
  Arms: Refined grain rice

SUMMARY:
Food products derived from cereal grains constitute a major part of the daily diet of many Americans . For example, a typical Chinese American eats rice about 9.5 times a week on an average. However, most of these foods are derived from refined grain. During the refining process grains are stripped of their bran and germ which results in depletion of several biologically active constituents including fiber, anti-oxidants, phytoestrogens and minerals. From observational studies there is evidence for a protective effect of whole-grain foods with regard to the development of type 2 diabetes. More recently, higher intake of whole grains was also associated with decreases in insulin resistance - a risk factor related to the development of type 2 diabetes.

In this randomized study the investigators plan to replicate this beneficial effect of improving insulin sensitivity in patients with pre-diabetes and go a step further by exploring the potential mechanisms by which this benefit may occur. The investigators will assess the effect of consuming a whole-grain-rich diet on levels of advanced glycation endproducts (AGE), RAGE (receptor for AGE) and markers of inflammation and oxidative stress - all of which have been shown to play an important role in the pathogenesis of diabetes mellitus. The investigators will also look for correlations between the levels of these markers with insulin sensitivity to identify potential mechanisms of pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years to unlimited, both genders.
2. At least one meal per day included rice in the seven days prior to enrolment.
3. No current diagnosis of Diabetes Mellitus (DM).
4. Fasting blood glucose value between 100 to 125 mg/dl and/or Hemoglobin A1c levels between 5.7%-6.4%.
5. ≥ 2 visits with primary care physician to establish compliance

Exclusion Criteria:

1. Special diets (e.g. vegetarian)
2. Use of medications that would affect blood sugar levels (e.g. steroids)
3. Allergy to any type of grain
4. Body weight fluctuation over the past 180 days of ≥ 10%
5. Planning to significantly change level of physical activity during the time of study.
6. Planning to move out of town or take a vacation for ≥ 14 days during the time of the study
7. Current smoker
8. Consumption of greater than 2 alcoholic drinks per day
9. History of malignancy and overt cardiovascular disease (apart from hypertension).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Homeostatic Model Assessment (HOMA) Index | 0
  Estimates insulin resistance and β-cell function from fasting glucose and insulin levels
Homeostatic model assessment(HOMA) index | 6 weeks
  Estimates insulin resistance and β-cell function from fasting glucose and insulin levels
Homeostatic model assessment (HOMA) index. | 12 weeks
  Estimates insulin resistance and β-cell function from fasting glucose and insulin levels

SECONDARY OUTCOMES:
Carboxymethyl lysine (CML) | 0, 6 and 12 weeks
  Advanced glycation end product (in blood and urine)
Methylglyoxal (MG) | 0, 6 and 12 weeks
  Advanced glycation end product (in blood and urine)
IL-6 | 0, 6 and 12 weeks
  Inflammatory marker
Receptor for advanced glycation endproducts (RAGE) | 0, 6 and 12 weeks
  Receptor for advanced glycation endproducts
Sirtuin 1 | 0, 6 and 12 weeks
  A protein that in humans is encoded by the SIRT1 gene and regulates processes such as apoptosis and muscle differentiation by deacetylating key proteins. It is down regulated in cells that have high insulin resistance and inducing its expression increases insulin sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Uribarri, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] McKeown NM, Meigs JB, Liu S, Wilson PW, Jacques PF. Whole-grain intake is favorably associated with metabolic risk factors for type 2 diabetes and cardiovascular disease in the Framingham Offspring Study. Am J Clin Nutr. 2002 Aug;76(2):390-8. doi: 10.1093/ajcn/76.2.390. PMID 12145012
- [Background] Fung TT, Hu FB, Pereira MA, Liu S, Stampfer MJ, Colditz GA, Willett WC. Whole-grain intake and the risk of type 2 diabetes: a prospective study in men. Am J Clin Nutr. 2002 Sep;76(3):535-40. doi: 10.1093/ajcn/76.3.535. PMID 12197996
- [Background] Montonen J, Knekt P, Jarvinen R, Aromaa A, Reunanen A. Whole-grain and fiber intake and the incidence of type 2 diabetes. Am J Clin Nutr. 2003 Mar;77(3):622-9. doi: 10.1093/ajcn/77.3.622. PMID 12600852
- [Background] Liese AD, Roach AK, Sparks KC, Marquart L, D'Agostino RB Jr, Mayer-Davis EJ. Whole-grain intake and insulin sensitivity: the Insulin Resistance Atherosclerosis Study. Am J Clin Nutr. 2003 Nov;78(5):965-71. doi: 10.1093/ajcn/78.5.965. PMID 14594783
- [Background] Steffen LM, Jacobs DR Jr, Murtaugh MA, Moran A, Steinberger J, Hong CP, Sinaiko AR. Whole grain intake is associated with lower body mass and greater insulin sensitivity among adolescents. Am J Epidemiol. 2003 Aug 1;158(3):243-50. doi: 10.1093/aje/kwg146. PMID 12882946